CLINICAL TRIAL: NCT06727227
Title: REal-world Study of Trastuzumab deruXtecan in Patients With unresectabLe or Metastatic Breast Cancer Expressing HER2-lOw From BulgaRia and SlovEnia (EXPLORE)
Brief Title: Real-world Study of Trastuzumab Deruxtecan in Patients With Unresectable or Metastatic HER2-low Breast Cancer
Acronym: EXPLORE
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9673R00055
Record Dates: First submitted 2024-11-20; First posted 2024-12-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: trastuzumab deruxtecan — T-DXd

SUMMARY:
A longitudinal, non-interventional study with trastuzumab deruxtecan for patients with HER2-low expressing unresectable or metastatic breast cancer in Bulgaria and Slovenia

DETAILED DESCRIPTION:
EXPLORE Non-Interventional Study for HER2-low Breast Cancer Treatment with T-DXd

Background:

HER2 is a prognostic marker in various cancers, including breast cancer (BC). Traditionally categorized as HER2-positive or HER2-negative, recent advancements with anti-HER2 ADCs, like trastuzumab deruxtecan (T-DXd), have shown benefits for HER2-low status BC. The DB-04 trial demonstrated significant survival benefits with T-DXd, leading to its EMA approval for HER2-low BC in January 2023.

Study Rationale:

Limited real-world evidence exists for T-DXd in HER2-low BC, particularly in the Balkans. The EXPLORE study aims to fill this gap by collecting real-world data in Bulgaria and Slovenia.

Objectives:

Primary Objective:

Describe real-world Time to Next Treatment (rwTTNT1) of T-DXd in HER2-low unresectable or metastatic BC (mBC).

Secondary Objectives:

Describe pre-T-DXd treatment patterns at baseline. Describe patient demographics and clinical characteristics at baseline. Describe rwTTNT1 by prior therapy lines in the metastatic setting and by hormone receptor (HR) status.

Evaluate real-world Time to Treatment Discontinuation (rwTTD1).

Exploratory Objectives:

Evaluate real-world progression-free survival (rwPFS1). Characterize subsequent treatments and post-progression endpoints (rwTTNT2, rwTTD2, rwPFS2).

Describe biopsy patterns. Evaluate reasons for discontinuation (rwTTNT1 and rwTTNT2). Describe T-DXd treatment changes over time. No formal hypothesis is set.

Methods:

Study Design:

Observational, longitudinal, non-interventional study in Bulgaria and Slovenia. Patients with unresectable or mBC starting T-DXd within 30 days of enrolment. Data from hospital charts at routine visits.

Population:

Adults (≥18 years) with HER2-low mBC, initiating T-DXd independent of the study.

Exposure:

T-DXd treatment details (dose, duration) and other therapies recorded. Recommended T-DXd dose: 5.4 mg/kg IV every 3 weeks.

Outcomes:

Primary: Time from T-DXd initiation to subsequent therapy or death. Exploratory: Various survival measures, biopsy patterns, reasons for discontinuation, and treatment changes.

Sample Size:

Approximately 135 patients (100 in Bulgaria, 35 in Slovenia).

Statistical Analysis:

Descriptive analyses for cohort characteristics. Kaplan-Meier method for time-to-event endpoints. Subgroup analyses by prior therapy lines and HR status.

Data Collection:

Data from paper or electronic health records. Single anonymized dataset via electronic case report forms (CRFs).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥18 years) with histological or cytological confirmed diagnosis of unresectable or mBC.
* Documented HER2-low status (IHC1+, IHC2+/ISH-) in patients who have received prior chemotherapy in the metastatic setting or documented HER2-low status (IHC 1+, IHC 2+/ISH-) in patients who have developed disease recurrence during or within 6 months of completing adjuvant chemotherapy.
* Recent prior decision to initiate therapy of T-DXd per SmPC (up to 30 days). Documentation confirming this decision will be required and collected.
* Able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* History of other primary malignancies in 2 years prior to unresectable or mBC diagnosis.
* Patients who at time of data collection for this study are participating in or have participated in an interventional study that remains blinded.
* HER2-low status patients who have previously documented HER2+ status in the same tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population:
  Criteria:
  Age: Adult patients (≥18 years). Diagnosis: Confirmed diagnosis of unresectable or metastatic breast cancer (mBC).
  HER2 Status: Documented HER2-low status. Treatment Decision: Patients for whom the decision to initiate trastuzumab deruxtecan (T-DXd) treatment has been made independently and prior to enrolment in the study.
  Enrollment:
  Timing: Patients must be enrolled within 30 days before the administration of the first T-DXd infusion.
  Consent: Patients must provide written informed consent for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Real-world Time to Next Treatment (rwTTNT1, median, 95% CI, measured in months) | Baseline up to 19 months
  The duration from initiation of trastuzumab deruxtecan (T-DXd) treatment to the start of the subsequent therapy or death from any cause, whichever occurs first, assessed up to 19 months.

SECONDARY OUTCOMES:
Describe type and proportion of previous treatments for unresectable or mBC and comorbidities | Baseline
  Prior treatments: surgery, chemotherapy, radiotherapy, therapies in neoadjuvant/adjuvant/advanced setting; treatment line (special focus should be given on endocrine and chemotherapy recycling in the metastatic setting). The timeline for these treatments will include all therapies administered from the time of breast cancer diagnosis.
Duration of previous treatments and number of treatment lines | Baseline
  Start and stop date, if available
Response to previous treatments | Baseline
  To describe patients' response to previous treatment, as applicable: clinical response (partial response/complete response/stable disease/disease progression; if progression: date and site of progression)
Mean (SD) age at diagnosis | Baseline
  Describe the patients' mean (SD) age at diagnosis
Mean (SD) age at T-DXd start | Baseline
  To describe patients' mean (SD) age at T-DXd start
Proportion of males and females | Baseline
  To describe the proportion of males and females
Proportion of patients with HR+ vs HR- tumors | Baseline
  Describe the proportion of patients with HR+ vs HR- tumors
Distribution by smoking status | Baseline
  Describe the patients' smoking status. Includes electronic cigarettes/vapes
Type and proportion of comorbidities | Baseline
  Comorbidities (including cardiovascular diseases, pulmonary disorders, hepatic disorders, renal disorders, blood and lymphatic system disorders, metabolism and nutrition disorders, gastrointestinal disorders, hepatobiliary disorders, central nervous system [CNS] disorders, eye disorders, skin disorders and musculoskeletal and connective tissue disorders, infections and infestations and other relevant
Distribution by ECOG status | Baseline
  Describe patients' ECOG PS at index date
mean (SD) duration of disease (at index), measured in months or years | Baseline
  Describe patients' mean duration of disease through date of initial diagnosis and date of diagnosis of unresectable or metastatic breast cancer, as applicable
HER2-low status and type and proportion of metastatic sites | Baseline
  Describe patients' HER2-low status and type and proportion of metastatic sites through most recent HER2-low status, new metastatic sites since the time of mBC diagnosis, disease burden (all disease sites, including the presence/absence of brain metastases [stable/active]
rwTTNT1 by Number of Prior of Therapy Lines for Metastatic Disease (median, 95% CI, measured in months, 1 vs 2 vs 3+ Lines) | Baseline up to 19 months
  Describe rwTTNT1 stratified by the number of prior therapy lines in the metastatic setting.
rwTTNT1 by HR-status (median, 95% CI, measured in months, HR+ vs HR-) | Baseline up to 19 months
  Describe rwTTNT1 stratified by hormone receptor (HR) status.
Real-world Time to Treatment Discontinuation (rwTTD1, median, 95% CI, measured in months) | Baseline up to 19 months
  Evaluate the duration from the start of T-DXd treatment until its discontinuation or death, whichever occurs first.

OTHER OUTCOMES:
Real-world Progression-Free Survival (rwPFS1, median, 95% CI, measured in months) | Baseline up to 19 months
  Evaluate the duration from the start of T-DXd treatment until disease progression or death, whichever occurs first.
Real-world Time to Second Next Treatment (rwTTNT2, median, 95% CI, in months) | Baseline up to 19 months
Real-world Time to Subsequent Treatment Discontinuation (rwTTD2, median, 95% CI, measured in months) | Baseline up to 19 months
Real-world progression free survival 2 (rwPFS2, median, 95% CI, measured in months) | Baseline up to 19 months
Biopsy Patterns (number of biopsies conducted prior to the start of T-DXd treatment) | Baseline, assessed for the past 10 years
  Describe the number of biopsies conducted prior to the start of T-DXd treatment.
Biopsy Patterns (the time from the last fresh biopsy to the start of T-DXd treatment, measured in months or years) | Baseline, assessed for the past 10 years
  Describe the time from the last fresh biopsy to the start of T-DXd treatment.
Reasons for Discontinuation (rwTTNT1 and rwTTNT2) | Baseline up to 19 months
  Evaluate the reasons for discontinuation of T-DXd treatment and subsequent therapy due to disease progression, adverse events, or other reasons.
T-DXd Treatment Changes Over Time | Baseline up to 19 months
  Proportion of patients with dose changes, proportion of patients with dose reductions, interruption(s), or treatment discontinuation

CONTACTS AND LOCATIONS:
Locations (8):
- Bulgaria (6):
  - Research Site, Panagyurishte, Pazardzhik
  - Research Site, Burgas
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
- Slovenia (2):
  - Research Site, Ljubljana
  - Research Site, Maribor

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/